CLINICAL TRIAL: NCT00257725
Title: Long-Duration Stimulant Treatment of ADHD in Young Children-Feasibility Study
Brief Title: Long-Duration Stimulant Treatment Study of ADHD in Young Children
Acronym: B-MPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Laurence Greenhill, Research Psychiatrist 2, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4939
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Attention-deficit/hyperactivity disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADHD Treatment Group (Experimental): Single-arm, open-label, once-daily-dosing of long-duration beaded MPH (B-MPH) at 10-30 mg (flexible titration) in 4-to-5 year old children with ADHD.
  Interventions: Drug: B-MPH

INTERVENTIONS:
Drug: B-MPH — Dosage form is a 20 mg capsule to be given once daily in the morning for 30 days
  Other Names: Ritalin LA

SUMMARY:
This study will evaluate if Ritalin LA™ is safe and effective for ADHD treatment in 4-to-5-year olds.

DETAILED DESCRIPTION:
This is a single site, open-label, four-week feasibility study of long-duration beaded methylphenidate (B-MPH), also known as Ritalin LA™. B-MPH is a FDA-approved medication for children 6 years and older with attention-deficit/hyperactivity disorder (ADHD), but there are no studies of its use in preschoolers. This study will evaluate the safety and effectiveness of B-MPH for ADHD treatment in 4-to-5-year old children.

Total study duration is approximately 5 weeks. It includes a screening evaluation and 4 weeks of B-MPH treatment with doses ranging from 10 to 30 mg (based on the individual tolerability and efficacy). The study doctor will conduct parent-training sessions during the treatment visits.

ELIGIBILITY:
Inclusion Criteria:

1. Parents/guardians and children must speak English and/or Spanish; parents/guardians must sign consent form; children must verbally assent.
2. Boys and girls from 4-5 years old (inclusive) at screening.
3. Children who meet the DSM-IV criteria for a primary diagnosis of ADHD (combined or hyperactive subtype), with symptoms present for at least 9 months.
4. Children who demonstrate adequate need for treatment due to ADHD symptom-severity and clinical impairment.
5. Children with IQ of at least 70 confirmed by valid IQ test.
6. Children who are in educational settings (pre-school, kindergarten, or elementary school program) with at least 8 same-age peers for at least two half days weekly.
7. Parents and children who can attend weekly study visits.
8. Children who are naïve to ADHD medications; received ADHD medications in the past but are not currently treated; or on ADHD medications but finding them inconvenient (due to short duration of action) or not very helpful

Exclusion Criteria:

1. Children and parents/guardians who do not understand or cannot follow necessary instructions; children and parents who are unwilling to comply with study procedures or cooperate with child psychiatrist.
2. Children taking excluded medications.
3. Children with history of intolerance to MPH/stimulant medications or no response to adequate stimulant trials.
4. Children with current adjustment disorder, autism, psychosis, bipolar disorder, significant suicidality, or other psychiatric disorders.
5. Children with history of physical, sexual, or emotional abuse, which lead to a significant impact on the clinical presentation and potentially some ADHD symptoms.
6. Children with screening abnormalities deemed clinically significant by child psychiatrist.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2005-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence L Greenhill, MD, Principal Investigator — New York State Psychiatric Insitute
Locations (1):
- New York State Psychiatric Insitute, New York, New York, United States

REFERENCES:
- [Result] Maayan L, Paykina N, Fried J, Strauss T, Gugga SS, Greenhill L. The open-label treatment of attention-deficit/hyperactivity disorder in 4- and 5-year-old children with beaded methylphenidate. J Child Adolesc Psychopharmacol. 2009 Apr;19(2):147-53. doi: 10.1089/cap.2008.053. PMID 19374023

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through the NYSPI Child and Adolescent Evaluation Service (CAPES), physician referrals, local and web advertising, and flyers. Recruitment took place between March 2005 and August 2007
Pre-assignment Details: The study included screening and one-week washout (if needed). All participants were entered into the study without incident.
Period: Overall Study
Arm/Group | ADHD Treatment Group
Started | 11
Completed | 8
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Groups:
- Single-arm Open-label B-MPH Treatment in Preschoolers w ADHD: Single-arm, open-label, once-daily-dosing of long-duration beaded MPH (B-MPH) at 10-30 mg (flexible titration) in 4-to-5 year old children with ADHD.
Arm/Group | Single-arm Open-label B-MPH Treatment in Preschoolers w ADHD
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.1 (.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Swanson, Nolan, and Pelham Questionnaire (SNAP-IV)
Description: The SNAP-IV Rating Scale is a revision of the Swanson, Nolan and Pelham (SNAP) Questionnaire (Swanson et al, 1983). The SNAP-IV is based on a 0 to 3 rating scale: Not at All = 0, Just A Little = 1, Quite A Bit = 2, and Very Much = 3. Subscale scores on the SNAP-IV are calculated by summing the scores on the items in the subset and dividing by the number of items in the subset. The score for any subset is expressed as the Average Rating-Per-Item, as shown for ratings on the ADHD-Inattentive (ADHD-I) subset.
  Sub scale ranges from 0-3. Higher scores mean better outcome. Change score from baseline is reported.
Time Frame: week 5
Population: Intent to treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ADHD Treatment Group
Number analyzed (Participants) | 11
score on a scale | -1.09 (0.73)
Statistical Analysis 1: Comparison: ADHD Treatment Group; Test type: Superiority or Other; p = 0.01, paired t-test; Mean Difference (Net) = -1.09, Standard Deviation 0.73

2. Primary Outcome: Clinical Global Impressions-Severity (CGI-S)
Description: CGI-S is designed to assess severity of illness on a seven-point scale: 1 = normal (not at ll ill) to 7 = among the most extremely ill patients.
  Range: 0-7, higher score means worse outcome. Change from baseline is reported.
Time Frame: week 5
Population: intent to treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ADHD Treatment Group
Number analyzed (Participants) | 11
score on a scale | -1.64 (1.29)
Statistical Analysis 1: Comparison: ADHD Treatment Group; Test type: Superiority or Other; p = 0.01, paired t-test; Mean Difference (Net) = -1.64, Standard Deviation 1.29

3. Primary Outcome: Children's Global Assessment Scale (C-GAS)
Description: Children's Global Assessment Scale (C-GAS) is designed to assess overall functioning across settings. The scale is rated from 1 to 100, with lower scores reflecting poorer adjustment. Change from baseline is reported.
Time Frame: week 5
Population: intent to treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ADHD Treatment Group
Number analyzed (Participants) | 11
score on a scale | 10.55 (7.70)
Statistical Analysis 1: Comparison: ADHD Treatment Group; Test type: Superiority or Other; p = 0.01, paired t-test; Mean Difference (Net) = 10.55, Standard Deviation 7.70

ADVERSE EVENTS:
Time Frame: 5 weeks (Baseline and 4 treatment visits)
Description: Using open-ended questions, the child psychiatrist elicited information about adverse events at baseline and at each subsequent visit. Information was obtained by observation and direct questioning such as, "Have you had any (other) medical problems since your last visit?" or "Have you felt different in any way since your last visit?"
Arm/Group | Single-arm Open-label B-MPH Treatment in Preschoolers w ADHD
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Single-arm Open-label B-MPH Treatment in Preschoolers w ADHD (N=11)
Decreased Appetite (Metabolism and nutrition disorders) | 7
Gastrointestinal Pain (Gastrointestinal disorders) | 2
Emotional Lability (Psychiatric disorders) | 2
Trouble Sleeping (Nervous system disorders) | 3
Sedation (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Increased Sensitivity (Nervous system disorders) | 1
Eye Twitching (Nervous system disorders) | 1/1
Headache (Nervous system disorders) | 1
Fever (General disorders) | 1
Virus with fever and headache (General disorders) | 1
Nasal Congestion (General disorders) | 1
Eye Redness (General disorders) | 1

LIMITATIONS AND CAVEATS:
The conclusions of this study are limited by its small size, the open-label design, and the possible confound of the parent training intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes